CLINICAL TRIAL: NCT05078567
Title: An Open Labeled Exploratory Study to Evaluate the Application of Natural Lactic Acid Enriched Cream in Adults With Plaque Psoriasis
Brief Title: Exploratory Study to Evaluate the Application of NLAC Cream in Adults With Plaque Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLACCLAS02
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm open label study (Experimental): Topical used natural lactic acid-enriched cream twice daily.
  Interventions: Device: 5% Natural Lactic Acid-enriched Cream

INTERVENTIONS:
Device: 5% Natural Lactic Acid-enriched Cream — The subjects were required to topically apply natural lactic acid-enriched cream twice daily in the morning and evening for the treatment duration of 12 weeks.

SUMMARY:
Psoriasis is a chronic and immune mediated skin disorder that presents with plaques of thickened, scaly skin. Up to 71% patients suffer from psoriasis, leading to high impact on their daily life. Plaque psoriasis is the most common type which causes thick, scaly patches of skin. Although the treatment of moderate-to-severe psoriasis has been improved with the new launched biologics, topical therapies continue to play a key role in the management of mild-to-moderate psoriasis. Up to 80% of patients of psoriasis use topical agents as their first-line therapy, including topical vitamin D analogs, corticosteroids, vitamin A analogs, and anthralin. There are well-documented concerns and limitations with current topical treatments. In this study, we propose a nature lactic acid enriched cream with a high safety profile as an alternative choice for patients with plaque psoriasis. Lactic acid is a natural moisturizing factor, which exists in healthy skin. It can efficiently prevent water loss from the skin and alleviate allergic reactions caused by dry skin. The moisturized function of lactic acid has made it became a commonly used additive in a wide variety of skincare products, such as lotion, cream, butter and spray. This product is rich in natural lactic acid generated by the fermentation of probiotics, and therefore can relieve skin itching caused by skin dryness, and resume the water-holding capability of the skin by removing abnormally proliferative stratum corneum as well as inducing collagen production. Importantly, this product is a steroid-free product with safety and without any induced adverse effects in use. This product is also can be a promising option other than steroids to be applied for the mitigation of recurrent symptoms in plaque psoriasis by resuming the water-retention ability of skin and rebuilding skin barrier function.

DETAILED DESCRIPTION:
I. Study Purpose

- Hypothesis: Natural lactic acid-enriched cream improves the Psoriasis Area and Severity Index scores in plaque psoriasis patients.

- Primary Objective: To assess the clinical efficacy of natural lactic acid-enriched cream for the proportion of subjects who achieve a Physician Global Assessment (PGA) score of clear (0) or almost clear (1) with a minimum 2-grade improvement from Baseline in patients with plaque psoriasis.

* Secondary Objectives:

  1. To assess the safety of 12 week-treatment of natural lactic acid-enriched cream application, as determined by the count of serious and non-serious treatment-emergent adverse events (AEs) during the study period.
  2. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with plaque psoriasis.
  3. To assess the TEWL, transepidermal water loss of natural lactic acid-enriched cream.

     II. Study Design and Methodology
* Subject This is an open-labeled exploratory study to evaluate safety and efficacy of natural lactic acid-enriched cream in adults with plaque psoriasis. The study was conducted at one medical center in Taiwan.
* Sample size:

Approximately 10 subjects who meet the criteria for study enrollment, will be treated with natural lactic acid-enriched cream.

- Treatment duration: The subjects were required to topically apply natural lactic acid-enriched cream twice daily in the morning and evening for the treatment duration of 12 weeks.

The study includes 3 periods: screening (up to 4 weeks), treatment (12 weeks), and post-treatment follow-up (4 weeks). Study visits occur at screening; at weeks 1, 2, 4, 8 and 12; and 2 and 4 weeks after the completion of treatment (weeks 14 and 16). The study will be conducted in the Department of Dermatology, Taipei Medical School Shuang Ho Hospital, Ministry of Health and Welfare.

- Investigational Product (IP) Natural lactic acid enriched cream: The natural lactic acid enriched cream was produced by Microbio Co. Ltd. and contained active ingredient 5% lactic acid is listed at 7 CFR Part 205.605 (a) as an approved nonsynthetic material produced by microbial fermentation.

* Inclusion Criteria:

  1. Male and female subjects ages 20 to 65 years with clinical diagnosis of chronic plaque psoriasis and stable disease for at least 6 months prior to the study.

  2. Capable of giving written informed consent 3. BSA involvement ≥ 5% and ≤ 10% 4. A PGA score of 3 (moderate) at screening and baseline 5. One target plaque located on the trunk or proximal parts of extremities (excluding knees, elbows, and intertriginous areas) that is at least 3 (centimeter) cm х 3 cm in size at Screening and Baseline with a severity representative of the subject's overall disease.

  6. Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study, including screening, during the treatment period, and for at least 4 weeks after the last exposure to study treatment
* Exclusion Criteria:

  1. Psoriasis other than plaque variant 2. Acute active bacterial, fungal, or viral (herpes simplex, herpes zoster, chicken pox) skin infection within 1 week prior to the Baseline visit; chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to the Baseline visit Significant dermatologic or inflammatory condition other than plaque psoriasis that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study 4. Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 4 weeks prior to the Baseline visit and/or plans to have such exposures during the study which could potentially impact the subject's psoriasis 5. Use of any prohibited medication within the indicated period before the first dose of study drug:

  -- Within a minimum of 5 half lives for biologic agents

  -- Within 4 weeks for systemic immunosuppressive or immunomodulating agents, fumaric acid derivatives, vitamin D3 and analogs, retinoids, psolarens, corticosteroids, adrenocorticotropic hormone analogs, and tazarotene
  * 2 weeks for immunizations with a live viral component
  * Drugs known to possibly worsen psoriasis, unless on a stable dose for > 12 weeks
  * With the exception of non medicated emollients, 1 week for topical treatments including corticosteroids, immunomodulators, anthralin (dithranol), vitamin D derivatives or coal tar
  * Any investigational product within 30 days, 5 half lives, or twice the duration of the biological effect of the study drug (whichever is longer) prior to first dose of study drug 6. Pregnant females or lactating females 7. Subjects have an allergic history of soybean and soybean derivatives. 8. History of sensitivity to the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates the subject's participation in the study
* Primary Endpoint:

Numbers of subjects who achieve a Physician Global Assessment (PGA) score of clear (0) or almost clear (1) with a minimum 2 grade improvement from Baseline at Week 12

- Secondary Endpoints:

1. Number of subjects with ≥ 75% improvement in Psoriasis Area and Severity Index (PASI) from Baseline at Week 4, 8 and 12.
2. Number of subjects with a PGA score of 0 or 1 at Week 4, 8, and 12.
3. Mean change in percent of total body surface area (%BSA) affected from Baseline to at Week 4, 8 and 12.
4. Number of subjects with ≥90% improvement in PASI score from Baseline to Week 4, 8 and 12.
5. Mean Change in PASI Score From Baseline to Week 4, 8 and 12.
6. Mean Change in PGA Score From Baseline to Week 4, 8 and 12.
7. The mean percentage change from baseline in trans epidermal water loss (TEWL) to Week 4, 8 and 12.

   - Safety Endpoint: The incidence of adverse events.

   - Experimental Groups: single arm, natural lactic acid enriched cream Clinical sample collection: To explore the diversity of the skin microbiome, skin microbiota will be harvested by swapping method at day 1 baseline visit, weeks 4, 12 and 16. DNA sequencing will be applied to clarify the composition of cutaneous microbiota at indicated time points.

   III. Statistical Analysis - General Statistics: For continuous variables, the following will be presented: mean, median, standard deviation, minimum and maximum. The comparison between two treatment groups and the comparison within group will be tested by using two independent t-test and paired t-test, respectively. If the normal assumption is violated, the Wilcoxon rank-sum and Wilcoxon signed-rank test will be conducted, respectively.

   For categorical variables, the numbers and percentages of subjects will be listed and summarized. Comparison for percentages will be performed using the Chi-square test and McNemar's test when comparing results in the same patient. The Fisher's exact test will replace the Chi-square test when any counting of the expected frequency is less than 5.

   - Endpoints: To perform the primary efficacy and other endpoints for continuous variable, two independent t-test will be used. If the normal assumption is violated, the non-parametric method of Wilcoxon rank-sum test will be applied for analysis. Significant level will be adopted with two-side at 0.05.

   For categorical variables, the Chi square test will be used. When any counting of the expected frequency is less than 5, the Fisher's exact test will be conducted. Significant alpha level will be adopted at 0.05

   - Safety: Adverse events will be coded by preferred term (PT) and system organ class (SOC) by the latest version of MedDRA. Adverse events will be summarized by severity, relationship to study drug, SAEs, and AEs leading to discontinuation of study drug.

   Physical examination findings will be presented in a tabulated listing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ages 20 to 65 years with clinical diagnosis of chronic plaque psoriasis and stable disease for at least 6 months prior to the study.
2. Capable of giving written informed consent
3. BSA involvement ≥ 5% and ≤ 10%
4. A PGA score of 3 (moderate) at screening and baseline
5. One target plaque located on the trunk or proximal parts of extremities (excluding knees, elbows, and intertriginous areas) that is at least 3 (centimeter) cm х 3 cm in size at Screening and Baseline with a severity representative of the subject's overall disease.
6. Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study, including screening, during the treatment period, and for at least 4 weeks after the last exposure to study treatment

Exclusion Criteria:

1. Psoriasis other than plaque variant
2. Acute active bacterial, fungal, or viral (herpes simplex, herpes zoster, chicken pox) skin infection within 1 week prior to the Baseline visit; chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to the Baseline visit
3. Significant dermatologic or inflammatory condition other than plaque psoriasis that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
4. Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 4 weeks prior to the Baseline visit and/or plans to have such exposures during the study which could potentially impact the subject's psoriasis
5. Use of any prohibited medication within the indicated period before the first dose of study drug:

   * Within a minimum of 5 half lives for biologic agents
   * Within 4 weeks for systemic immunosuppressive or immunomodulating agents, fumaric acid derivatives, vitamin D3 and analogs, retinoids, psolarens, corticosteroids, adrenocorticotropic hormone analogs, and tazarotene
   * 2 weeks for immunizations with a live viral component
   * Drugs known to possibly worsen psoriasis, unless on a stable dose for > 12 weeks
   * With the exception of non medicated emollients, 1 week for topical treatments including corticosteroids, immunomodulators, anthralin (dithranol), vitamin D derivatives or coal tar
   * Any investigational product within 30 days, 5 half lives, or twice the duration of the biological effect of the study drug (whichever is longer) prior to first dose of study drug
6. Pregnant females or lactating females
7. Subjects have an allergic history of soybean and soybean derivatives.
8. History of sensitivity to the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates the subject's participation in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Physician Global Assessment (PGA) score | Week 12
  Numbers of subjects who achieve a Physician Global Assessment (PGA) score of clear (0) or almost clear (1) with a minimum 2 grade improvement from Baseline at Week 12